CLINICAL TRIAL: NCT01274325
Title: Comparison of Anti-inflammatory Effects of Seroflo 125 Inhaler With Seretide Evohaler(25/125) in Patients With Asthma
Brief Title: Comparison of Anti-inflammatory Effects of Seroflo and Seretide in Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: si446/2010
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sereflo (Experimental): Sereflo (25/125)
  Interventions: Drug: Sereflo
- Seretide (Active Comparator): Seretide (25/125)
  Interventions: Drug: Seretide

INTERVENTIONS:
Drug: Sereflo — Patients take sereflo (25/125) 2 puffs twice a day for 4 weeks
  Arms: Sereflo
Drug: Seretide — Patients will take Seretide (25/125) 2 puffs twice a day for 4 weeks
  Arms: Seretide

SUMMARY:
The purpose of this study is to test hypothesis if Sereflo (ICS/LABA) could reduce airway inflammation in asthmatic patients in the same as Seretide.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 years
* Patients with asthma diagnosed by according to the American Thoracic Society criteria
* A baseline FEV1 > or = 50% predicted with a reversibility of FEV1 after therapy with inhaled salbuterol (2.5 mg) of FEV1 12% or with provocative concentration of a methacholine causing a 20% fall in FEV1 (PC20) of < or = 8 mg/mL
* Prescribed use of inhaled corticosteroids (any brand) for at least 12 weeks prior to study entry
* The daily prescribed dose of inhaled corticosteroids during the last 4 weeks prior to study entry should have been constant and at least 250 μg/day of fluticasone at least 400 μg/day of budesonide at least 500 μg/day of any other beclomethasone
* Be able to provide written informed consent

Exclusion Criteria:

* Any asthma exacerbation or respiratory tract infection affecting asthma within 4 weeks prior to the randomization visit
* Intake of oral, parenteral corticosteroids within 4 weeks and/or depot parenteral corticosteroid within 12 weeks prior to the randomization visits
* Current or previous smoker with a smoking history of > or = 10 pack years
* Previous randomization of treatment in the present study
* Known or suspected hypersensitivity to study therapy
* Use of any β-blocking agent, including eye-drops
* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive pill measures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophils | 4 weeks

SECONDARY OUTCOMES:
Exhaled nitric oxide | 4 weeks
Asthma control test scores | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong Maneechotesuwan, MD., PhD., Principal Investigator — Siriraj Hospital
Locations (2):
- Thailand (2):
  - Kittipong Maneechotesuwan, Bangkoknoi, Bangkok
  - Division of Respiratory Disease and TB, Siriraj Hospital, Bangkoknoi, BKK